CLINICAL TRIAL: NCT01683643
Title: Screening, Brief Intervention, and Referral to Treatment for Offenders
Acronym: SBIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michael Prendergast, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA031879 (NIH)
Record Dates: First submitted 2012-09-05; First posted 2012-09-12 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Substance Use; HIV Infections
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBIRT Group (Experimental): Baseline demographic data will be collected. Subjects will be screened for substance use risk using The Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) developed by the World Health Organization. Experimental subjects, in addition to their risk score and informational materials, will also receive a brief intervention and a referral to treatment appropriate to their risk score from trained health educators. The health educators will be provided by Homeless Health Care, Los Angeles.
  Interventions: Behavioral: SBIRT
- Control Group (Active Comparator): Baseline demographic data will be collected. Subjects will be screened for substance use risk using The Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) developed by the World Health Organization. Control subjects will receive only their risk score and informational materials regarding the health risks of substance use.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: SBIRT — Screening, brief intervention, and referral to treatment.
  Arms: SBIRT Group
Behavioral: Control Group — Control subjects will receive only their risk score and informational materials regarding the health risks of substance use.
  Arms: Control Group

SUMMARY:
The purpose of the study is to determine whether SBIRT is an effective intervention with inmates and to estimate the costs of providing SBIRT to this population.

DETAILED DESCRIPTION:
Screening, Brief Intervention, and Referral to Treatment (SBIRT) is an evidence-based practice that has been found to be effective in reducing alcohol and illicit drug use, mainly among persons recruited in medical centers, primary care offices, emergency rooms, and colleges and universities. But SBIRT has the potential to be applicable to other populations that have, or that are at risk for, substance use problems. In particular, offenders have high prevalence of drug and alcohol use at varying levels of severity and often do not receive adequate intervention, either because of limited availability of programs, low motivation, or lack of awareness of the consequences of their substance use.

The scientific aims of the study are:

1. Assess the effectiveness of SBIRT with offenders in terms of participation in brief intervention (if so indicated) and enrollment in treatment (if so indicated).
2. Assess the effectiveness of SBIRT with offenders in terms of drug use, criminal activity, and criminal justice involvement at 12 months following baseline.
3. Determine whether there are differences in acceptability, participation, and outcomes between men and women.
4. Determine the cost of providing the SBIRT intervention with this population.

The clinical aims of the study are:

1. To complement the use of SBIRT within Los Angeles County's substance abuse treatment system.
2. To expand prevention and treatment options for offenders with substance abuse problems.

To our knowledge, this would be the first rigorous test of SBIRT with an offender population.

We will recruit inmates at two Los Angeles County Sheriff jail facilities, one for men and one for women (25% of total sample), and randomly assign them to the treatment (SBIRT) group (N =400) or to the control (no intervention) group (N = 400). Baseline demographic data will be collected. Subjects in both groups will be screened for substance use risk using The Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) developed by the World Health Organization. Control subjects will receive only their risk score and informational materials regarding the health risks of substance use. Experimental subjects, in addition to their risk score and informational materials, will also receive a brief intervention and a referral to treatment appropriate to their risk score from trained health educators. The health educators will be provided by Homeless Health Care, Los Angeles. Twelve months after study admission, all study participants will be contacted for a follow-up interview. We will obtain records-based data on arrests and jail incarceration over the follow-up period from the Sheriff's Department and the California Department of Justice. We will also collect subject participation in publicly-funded treatment from the Substance Abuse Prevention and Control Division of the Los Angeles County Department of Health.

ELIGIBILITY:
Inclusion Criteria:

* The sample for the study will be drawn from an offender population who are within 2-3 weeks of their release from MCJ or CRDF in Los Angeles County. In addition, subjects must be:

  * At least 18 years of age
  * English or Spanish speaking
  * Not subject to extended jail or prison sentence
  * Able to provide informed consent to participate in the study

Exclusion Criteria:

* Study exclusion criteria:

  * Inability to provide informed consent to study participation because of cognitive impairment.
  * Inability to communicate in either English or Spanish
  * Refusal to complete Locator form for follow-up.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2012-04; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
A reduction in the use of drugs and alcohol | 12 months

SECONDARY OUTCOMES:
Participation in treatment | 12 months
Rearrest and incarceration | 12 months
Quality of life | 12 months
A reduction in HIV risk behaviors | 12 months
The cost benefit of SBIRT for offenders | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prendergast, Ph.D, Principal Investigator — UCLA Integrated Substance Abuse Programs; Jerry Cartier, M.A., Study Director — UCLA Integrated Substance Abuse Programs
Locations (1):
- University of California, Los Angeles, California, United States

REFERENCES:
- [Derived] Prendergast ML, McCollister K, Warda U. A randomized study of the use of screening, brief intervention, and referral to treatment (SBIRT) for drug and alcohol use with jail inmates. J Subst Abuse Treat. 2017 Mar;74:54-64. doi: 10.1016/j.jsat.2016.12.011. Epub 2016 Dec 30. PMID 28132701
- [Derived] Prendergast ML, Cartier JJ. Screening, brief intervention, and referral to treatment (SBIRT) for offenders: protocol for a pragmatic randomized trial. Addict Sci Clin Pract. 2013 Oct 23;8(1):16. doi: 10.1186/1940-0640-8-16. PMID 24499609